CLINICAL TRIAL: NCT03986099
Title: Community Based Virus Load Differentiated Care in Rural Africa
Brief Title: Community Based Antiretroviral Therapy (CBART) Among Children on Chronic ART
Acronym: CBART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biomedical Research and Training Institute, Zimbabwe (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: AP142/2017
Record Dates: First submitted 2019-03-27; First posted 2019-06-14 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: ART; HIV I Infection
Keywords: Children and adolescents; HIV therapy; Virologic suppression; Zimbabwe; Rural; GeneXpert; Point of care; SAMBA

STUDY DESIGN:
Intervention Model Description: Patients assigned to either point of care (POC) or standard of care (SOC)
Who Masked: Participant
Masking Description: Single blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): SOC viral load
- Near point of care (Active Comparator): POC viral load
  Interventions: Diagnostic Test: Monitoring virus load

INTERVENTIONS:
Diagnostic Test: Monitoring virus load — Near point of care
  Arms: Near point of care

SUMMARY:
A randomized, open label trial of two strategies for Virus Load Differentiated Care (VLDC) monitoring of virologic outcome in a rural community based treatment program in Zimbabwe.

DETAILED DESCRIPTION:
This is an open label randomized trial among HIV infected children and adolescents and young adults receiving ART at 8 treatment outreach sites near their homes provided by Chidamoyo Mission Hospital. The investigators will implement virus load (VL) testing at "near point of care" using either the GeneXpert Quant or the SAMBA to evaluate the safety, clinical and virologic outcomes of near POC monitoring of virus load at the Chidamoyo Christian Hospital in Mashonaland West Zimbabwe.

The investigators hypothesize that our proposed package of care will result in a decrease in virologic failure, increase virologic suppression and prevent drug resistance in this key population in a rural ART treatment program. Process and cost data will be collected for subsequent cost-analysis.

HIV infected children and adolescents on ART will be randomized (1:1) to either SOC (300) or a near POC VLDC monitoring. SOC VL is performed by Roche COBAS at the Provincial Hospital Chinhoyi and the results returned to the hospital within 4 weeks. Those randomized to near POC will be tested with the Cepheid GeneXpert assay and results are available within 3 days. Follow-up repeat testing for HIV RNA > 1,000 copies/ml is offered using the same virologic monitoring system at the next drug/clinic visit within 3 months.

The hypothesis is that viral load monitoring and potentially genotyping to sustain suppression to < 1,000 copies/ml will reduce treatment failure to < 15%. Secondary endpoints include the rate of drug switching and the evaluation and prevention of drug resistance. The study will enroll up to 600 children (3 -10) years and adolescents (11-21) years, providing data that will guide strategies for management of children and adolescents who are surviving on ART.

Primary Objective: To determine if implementation of point of care virus load differentiated care (POC virus load), targeted genotyping and mHealth tools will result in improved virologic suppression among children and adolescents (<21years) on ART.

Sample size: The primary study endpoint is viral load suppression at 48 weeks among PLWHA < 21 years old, using VLDC implemented as near POC compared to SOC semi- annual virus load testing. The investigators will enroll young PLWHA from eight communities and the Chidamoyo Hospital Clinic as a rolling prospective cohort. The investigators hypothesize that an intervention package of digitized data, local immediate POC Virus load and genotype will result in > 90% virologic suppression after 1 year. The estimated minimum sample size to detect at least a 15% increase in virologic suppression with 90% power, at significance level α=0.05 assuming 10% loss to follow up rate (LTFU) rate is 356 PLWHA on ART.

Secondary endpoints:

1. rate of switching from 1st to 2nd line.
2. frequency of Drug Resistance Mutations (DRM) among 1st and 2nd line virologic failures.
3. the frequency of Hepatitis B virus infection (HBSag).

In collaboration with Ben Gurion University Global Health, the investigators will perform an ethnographic survey over the course of the primary study. The objective is to develop formative research to understand the individual and community variation in suppression rate and drug switching including differences in virologic failure and adherence by age, gender, rural outreach site, orphan-hood/caregiver and socio-economic status.

ELIGIBILITY:
Inclusion Criteria:

- HIV positive children and adolescents on ART

Exclusion Criteria:

* Unable to consent
* Less than one year on ART

Ages: 2 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 451 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Viral load suppression | 48 weeks
  Viral load suppression

SECONDARY OUTCOMES:
Number of participants with confirmed virology failure who switched regimens | 96 weeks
  Change to second line regimen after confirmed virological failure
Drug resistance mutations | 96 weeks
  Provider initiated genotyping

CONTACTS AND LOCATIONS:
Overall Officials: Shungu Munyati, PhD, Principal Investigator — Biomedical Research and Training Institute
Locations (1):
- Chidamoyo Christian Hospital, Karoi, Mashonaland West, Zimbabwe

REFERENCES:
- [Derived] Kouamou V, Machekano R, Mapangisana T, Maposhere C, Mutetwa R, Manasa J, Shamu T, McCarty K, Munyati S, Mutsvangwa J, Bogoshi M, Israelski D, Katzenstein D. Clinic-based SAMBA-II vs centralized laboratory viral load assays among HIV-1 infected children, adolescents and young adults in rural Zimbabwe: A randomized controlled trial. PLoS One. 2023 Feb 14;18(2):e0281279. doi: 10.1371/journal.pone.0281279. eCollection 2023. PMID 36787296
- [Derived] Kouamou V, Machekano R, Mapangisana T, Maposhere C, Munyati S, Mutsvangwa J, Shamu T, McCarty K, Katzenstein D, Manasa J. Tenofovir, Lamivudine, and Dolutegravir Among Rural Adolescents in Zimbabwe: A Cautionary Tale. AIDS Res Hum Retroviruses. 2022 Oct;38(10):774-778. doi: 10.1089/AID.2021.0140. Epub 2022 Sep 7. PMID 35959737